CLINICAL TRIAL: NCT06236464
Title: Identification of the Pathogenetic Mechanisms Underlying Squamous Cell Carcinomas of the Anogenital Tract and of the Head-neck Region for the Development of Shared Therapeutic Strategies
Brief Title: Identification of the Pathogenetic Mechanisms Underlying Squamous Cell Carcinomas
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-MAD-2022-12376570; 9/23 oss (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma of the Anus
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Multiparameter analysis of each sample — Retrospective and prospective samples will be collected and analyzed for the study of molecular and viral biomarkers. Simultaneously, fibroblastic tumor-associated cells (CAFs) will be isolated from prospective samples. Through co-cultivation with immortalized cell lines derived from anogenital and head-neck SCCs, these CAFs will enable the production of 3D organoids for use in experiments assessing the response to telomerase and deacetylase SIRT1 inhibitors, both in vitro and in preclinical models.

SUMMARY:
This is a multicentric, retrospective, and prospective biomarker study.

DETAILED DESCRIPTION:
This is a multicentric, retrospective, and prospective biomarker study, involving a total of 170 patients with SCC (Squamous Cell Carcinoma) of the mucosa of the anogenital tract and head-neck region, recruited from INT-NA (n=50), UPO (n=40), AOUP (n=40), and ITB (n=40). Specifically, retrospective and prospective samples will be collected and analyzed for the study of molecular and viral biomarkers. Simultaneously, fibroblastic tumor-associated cells (CAFs) will be isolated from prospective samples. Through co-cultivation with immortalized cell lines derived from anogenital and head-neck SCCs, these CAFs will enable the production of 3D organoids for use in experiments assessing the response to telomerase and deacetylase SIRT1 inhibitors, both in vitro and in preclinical models.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 years, candidates for surgical treatment for squamous cell carcinoma of the anus, uterine cervix, vulva, and head-neck region (including microinvasive and invasive carcinomas) who are capable of understanding and willing to sign the informed consent form. Prospective patients must provide written informed consent before any procedures.

Exclusion Criteria:

Patients presenting any of the following criteria are not eligible for inclusion in this study. Exclusion criteria include:

1. Metastatic neoplasia
2. Treatment for other oncological pathologies
3. Congenital or acquired immunosuppression (HIV, organ transplant, pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with a histological diagnosis of squamous cell carcinoma (SCC) of the anus, cervix, vulva, oral cavity, and oropharynx. At least 170 cases of anal SCC (n=30), cervical SCC (n=30), vulvar SCC (n=30), oral cavity SCC (n=40), and oropharyngeal SCC (n=40) will be prospectively enrolled and retrospectively analyzed.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 30 months
  Identify shared molecular profiles in squamous cell carcinomas (SCC) of the mucosa of the anogenital tract and head-neck region, dependent on the presence of somatic mutations (e.g., TERT promoter mutations and viral HPV sequences).

SECONDARY OUTCOMES:
Secondary Endpoint | 30 months
  Inhibition of growth in organoids obtained from tumor cells mutated in the TERT promoter or expressing viral oncogenes and SIRT1.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lina Tornesello, M.D., Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (4):
- Italy (4):
  - Istituto Tumori IRCCS Giovanni Paolo II di Bari, Bari, Bari
  - Istituto Nazionale Tumori | "Fondazione Pascale", Napoli, Napoli
  - Università del Piemonte orientale, Novara, Novara
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Pisa

IPD SHARING:
Plan to Share IPD: No